CLINICAL TRIAL: NCT06704607
Title: Impact of Optimization of Nutritional State on the Outcome of Patients with Acute Exacerbation of Bronchiectasis
Brief Title: Optimization of Nutritional State on the Outcome of Patients with Acute Exacerbation of Bronchiectasis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, lecture of chest disease at assiut university, Assiut University
Other Study IDs: Bronchiectas nutritional state
Record Dates: First submitted 2024-10-27; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Bronchiectasis Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Bronchiectasis is a chronic respiratory condition characterized by the abnormal and permanent dilation of the bronchi, leading to recurrent respiratory infections, chronic cough, and significant morbidity. The disease has gained increasing recognition due to its rising prevalence and the substantial burden it places on healthcare systems .

Recent studies have highlighted the importance of nutritional status in managing chronic respiratory diseases, including bronchiectasis. Malnutrition is prevalent among patients with bronchiectasis, particularly those experiencing frequent exacerbations. It has been shown that underweight patients have lower lung function and may face worse clinical outcomes compared to those with normal weight . Specifically, a study found that underweight individuals had a significantly lower forced expiratory volume in one second (FEV1) compared to their normal-weight counterparts, indicating a direct correlation between nutritional status and respiratory function .

DETAILED DESCRIPTION:
To evaluate the effects of nutritional optimization on clinical outcomes in patients experiencing an acute exacerbation of bronchiectasis. Specifically, the study seeks to:

* Assess the Relationship Between Nutritional Status and Clinical Outcomes*: To investigate how improvements in nutritional status, measured through dietary intake, body weight, and biochemical markers, correlate with clinical outcomes such as length of hospital stay, frequency of exacerbations, and overall recovery.

  * *Evaluate the Effectiveness of Nutritional Interventions*: To determine the impact of specific nutritional interventions (e.g., high-protein diets, caloric supplementation, and micronutrient support) on the health status and recovery of patients during acute exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* *Age*: Adults aged 18 years and older.

  * Diagnosis*: Confirmed diagnosis of bronchiectasis, as established by clinical evaluation and imaging studies (e.g., chest CT scan).
  * Acute Exacerbation*: Patients presenting with acute exacerbation symptoms, such as increased sputum production, worsening dyspnea, or chest pain.
  * Nutritional Assessment*: Patients identified as malnourished or at risk of malnutrition based on the Subjective Global Assessment (SGA) or similar nutritional screening tools.

Exclusion Criteria:

* *Cognitive Impairment*: Patients with cognitive impairments that affect their ability to participate in the study or adhere to nutritional recommendations.

  * Current Enteral Feeding*: Patients receiving enteral nutrition or those with a feeding tube.

Recent Nutritional Interventions*: Patients who have recently undergone significant nutritional interventions (e.g., dietary changes, supplementation) within the past three months prior to enrollment.

*Pregnancy or Lactation*: Pregnant or lactating women, due to the need for specific nutritional considerations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Recruitment Patients will be recruited from inpatient wards. Informed consent will be obtained from all participants prior to enrollment.
  Nutritional Assessment
  * **Baseline Assessment**:
  * Nutritional status will be determined using the Subjective Global Assessment (SGA) and biochemical markers (e.g., serum albumin).
  * Dietary intake will be assessed using a 3-day food diary or 24-hour dietary recall method.
  * **Nutritional Optimization**: Patients identified as malnourished will receive a tailored nutritional intervention, which may include:
  * High-protein dietary recommendations.
  * Caloric supplementation through protein shakes or high-calorie snacks.
  * Micronutrient supplementation as need
  Data Collection
  Data will be collected at three time points:
  1. **Baseline**: Upon admission.
  2. **During Hospitalization**: After the implementation of nutritional interventions.
  3. **Follow-Up**: Six months post-discharge, assessing long-term outcomes.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Asses The Change In Quality of life | base line
  measured by the St. George's Respiratory Questionnaire (SGRQ).

REFERENCES:
- [Background] Martinez Garcia MA, Maiz Carro L, Catalan Serra P. [Treatment of non-cystic fibrosis bronchiectasis]. Arch Bronconeumol. 2011 Dec;47(12):599-609. doi: 10.1016/j.arbres.2011.06.003. Epub 2011 Jul 28. Spanish. PMID 21798654